CLINICAL TRIAL: NCT02952352
Title: A Culturally Tailored Intervention to Prevent Diabetes in American Indian Men
Brief Title: Nxstan: A Culturally Tailored Intervention to Prevent Diabetes in American Indian Men
Acronym: NARCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Odile Madesclaire, Senior Research Program and Operations Manager, Washington State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U261IHS0086-01-00
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Intervention (Experimental): Diabetes Prevention Program
  Interventions: Behavioral: Diabetes Prevention Program
- Delayed Intervention (Other): Diabetes Prevention Program
  Interventions: Behavioral: Diabetes Prevention Program

INTERVENTIONS:
Behavioral: Diabetes Prevention Program — Culturally adapted diabetes prevention program

SUMMARY:
To reduce modifiable diabetes risk factors' in overweight and obese AI men residing on the Colville reservation through a community-based, culturally informed intervention, the study specifically aims to: 1. conduct focus groups and interviews with adult members of Colville tribe to inform the adaptation, manualization and implementation of a culturally informed diabetes prevention program among overweight and obese AI men; 2. evaluate the effectiveness of a community-based, culturally informed diabetes prevention intervention by assessing between group changes.

DETAILED DESCRIPTION:
To reduce modifiable diabetes risk factors' in overweight and obese AI men residing on the Colville reservation through a community-based, culturally informed intervention, the study specifically aims to: 1. conduct focus groups and interviews with adult members of Colville tribe to inform the adaptation, manualization and implementation of a culturally informed diabetes prevention program among overweight and obese AI men; 2. evaluate the effectiveness of a community-based, culturally informed diabetes prevention intervention by assessing between group changes in: Primary Outcomes: weight, dietary fat and caloric intake, vegetable consumption, and physical activity; Secondary Outcomes: physical fitness, blood pressure, lipids, self-reported quality of life; and, 3. evaluate the sustainability of the diabetes prevention intervention by assessing participant perceptions of program component fit through focus group discussions with participants in the intervention and telephone interviews with those who left the program.

ELIGIBILITY:
Inclusion Criteria:

* Must be male and self-reported American Indian; Reside in or near Colville tribe; ages 21-65, A BMI ≥25 kg/m2 and/or a waist circumference >90 cm for men; no prior diabetes diagnosis; No history of heart disease, serious illness, cancer diagnosis in the last five years, or other conditions that may impede or prohibit participation; and, willingness to consent to randomization

Exclusion Criteria:

* Females, under 18 years old or older than 65 years

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Weight | 12 Weeks
  Percent weight loss

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure | 12 weeks
  blood pressure monitor
Stages of Change for weight loss | 12 weeks
  Transtheoretical model of stages of change questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Odile A Madesclaire, Principal Investigator — Washington State University
Locations (2):
- United States (2):
  - Confederated Tribes of the Colville Reservation, Nespelem, Washington
  - IREACH, Seattle, Washington